CLINICAL TRIAL: NCT03150654
Title: The Effect of Laser Pan-retinal Photocoagulation on Macular Pigment Optical Density in Cases With Diabetic Retinopathy
Brief Title: The Effect of Laser Treatment on Macular Pigment of Eye in Cases With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyon Kocatepe University Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2011-KAEK-2 2015/323
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Retinopathy; Retinal Degeneration; Macula Abnormality; Laser Burn of Retina
Keywords: macular pigment; macular pigment optical density; diabetic retinopathy; laser pan-retinal photocoagulation
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: sequential self-controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Laser pan-retinal photocoagulation (Experimental): Conventional laser pan-retinal photocoagulations were performed by using green laser photocoagulator, every month for 3 months
  Interventions: Device: Laser pan-retinal photocoagulation

INTERVENTIONS:
Device: Laser pan-retinal photocoagulation — Green laser photocoagulator
  Other Names: GYC-500 Vixi

SUMMARY:
It has been hypothesized that thermal damage of laser pan-retinal photocoagulation may affect macular pigment as well as inner layer cells in the retina, so it was aimed to investigate possible effect of conventional laser pan-retinal photocoagulation on macular pigment optical density in diabetic retinopathy patients without macular edema and pathology in this study.

DETAILED DESCRIPTION:
The local authorized clinical trials ethics committee approved the study and this study was performed following the principles of the Declaration of Helsinki (2008). Detailed information was given to patients about clinical applications and tests, and signed informed consent forms were also obtained from all patients. The 36 eyes of 36 patients, scheduled for laser pan-retinal photocoagulation treatment, with newly diagnosed proliferative diabetic retinopathy without macular edema or scarring between October 2015 - June 2016 were included in this sequential self-controlled clinical trial. Proliferative diabetic retinopathy was diagnosed with determination of neovascular proliferations is either on the disc (NVD) or elsewhere (NVE) except macular area in fundus examination with 90-diopter lens and fundus fluorescein angiography (FFA) (Heidelberg Spectralis, Heidelberg Engineering, Baden-Württemberg, Germany). Patients, detected macular fluid or edema by optical coherence tomography (OCT) (Cirrus HD 4000, Carl Zeis Meditec, CA, USA) in study eye, were excluded in the study. After providing information to patients about the disease and treatment; patients, predicted to show adherence to treatment, were enrolled in the study.

Ophthalmological examinations were performed in all cases. Firstly, visual acuity was recorded, and best-corrected visual acuity (BCVA) assessed using Snellen's chart and was converted to logarithm of the minimum angle of resolution (logMAR) for statistical analysis. After maximal pupil dilatation was achieved using 1% tropicamide and 10% phenylephrine eye drops, put once or twice, at ten minute intervals, slit-lamp examination was performed, and fundus was examined with 90-diopter indirect non-contact fundus lens, and ocular finds were recorded.

Prior to measurements the pupil was dilated to at least 7 mm diameter using a topical mydriatic agent. Macular pigment optical density (MPOD) levels were measured in the study eye using luminance differential thresholds test (MonPack System®, Metrovision, Perenchies, France), color perimetry technique at baseline before first PRP laser treatment and every month before laser treatment until the end of this study. The macular pigment absorbs blue light, and luminance differential thresholds test evaluates the density of the macular pigment by comparing the thresholds of perception of blue light and red light with a staircase technique similar to the technique used in automated perimetry. Luminance differential thresholds were measured for 2 stimuli: a blue stimulus (450-480 nm) absorbed by the MP, and a red one (615 nm) not absorbed. The stimuli were presented at the fovea and at 6 peripheral locations with an eccentricity of 3 to 10 degrees (0°, 0.8°, 1.8°, 2.8° and 3.8°, and the average of two measurements at 6.8° and 7.8° retinal eccentricity serves as the peripheral reference point). Tests parameters were Goldmann size III over a white background of 10 cd.m-2. The average values of the tested (decibel=dB) were converted to logarithm units (log unit) for statistical analysis (dB = 10log10 (Reference1/Reference2)). Because, decibel is always the comparison between two values. As a result, the decibel number is the same, although the measured power value is often different. Therefore, arithmetic operations with the numbers expressed in decibels would be inconvenient.

Conventional laser PRP treatments were performed under topical anesthesia by using green laser photocoagulator (GYC-500 Vixi® Nidek, Gamagori, Japan) and Volk® quadraspheric lens. PRP laser were applied in 300mW power, 200-400-500 μm spot size and 0.1-0.2 second pulse options, based upon preferences and comfort levels. When a pattern array was used, the spot separation was set at 0.5 times the burn width.

Laser parameters were evaluated based on a) area (A) (= πr2 × number of shots) r being the spot radius, which is half of the spot size (100-200-250 μm), and it was converted to square millimeters (mm2) for statistical analyses, b) treatment duration (t) (= 0.1 - 0.2 second × number of shots) and c) total energy (E) (= P × t) milijoules (mJ) P being the power, which is 300mW.

All examinations, MPOD and laser PRP parameters were repeated and recorded at 1st, 2nd, 3rd month before laser treatments and 6th month. Changes in the eating habits of patients were questioned at all study visits. All subjects were told to continue their normal diet, as no subjects were consuming supplements containing lutein or zeaxanthin.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity (BCVA) logMAR ≤0.4
* Newly diagnosis of PDR and initiation of conventional laser PRP treatment
* Between the ages of 40 and 65 years (40≤age≤65)

Exclusion Criteria:

* Corneal scarring, cataract or intravitreal hemorrhage that prevents appearance of the fundus
* Presence of macular pathologies such as AMD or choroidopathy
* Presence of macular edema or NVE in the macular area
* Detection of macular fluid or edema in OCT or FFA
* Previous laser PRP treatments
* Focal and / or grid photocoagulation requirements
* Previous refractive or vitreoretinal surgery
* Spherical refractive error ≥ ±6.00 D or cylinder refractive error ≥ ±3.00 D
* Systemic diseases that may affect the choroidal blood flow such as cardiological diseases
* Current use of carotenoid supplementation
* Changing eating habits
* Gastrointestinal diseases that could cause disturbance of dietary absorption

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
Change macular pigment optical density from baseline at 6 months | 1 month and 3 months
  Macular pigment optical density measures were repeated and recorded at 1st, 2nd, 3rd month before laser treatments and 6th month

SECONDARY OUTCOMES:
Correlation analysis between macular pigment optical density and panretinal laser photocoagulation parameters during 6 months | 6 months
  The correlations between macular pigment optical density outcomes and panretinal laser photocoagulation parameters (total energy, total area, total shots, total duration) were evaluated for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Dogan, Asst. Prof., Study Director — Afyon Kocatepe University Eye Clinics

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bone RA, Landrum JT, Friedes LM, Gomez CM, Kilburn MD, Menendez E, Vidal I, Wang W. Distribution of lutein and zeaxanthin stereoisomers in the human retina. Exp Eye Res. 1997 Feb;64(2):211-8. doi: 10.1006/exer.1996.0210. PMID 9176055
- [Background] Krinsky NI, Landrum JT, Bone RA. Biologic mechanisms of the protective role of lutein and zeaxanthin in the eye. Annu Rev Nutr. 2003;23:171-201. doi: 10.1146/annurev.nutr.23.011702.073307. Epub 2003 Feb 27. PMID 12626691
- [Background] Krinsky NI, Johnson EJ. Carotenoid actions and their relation to health and disease. Mol Aspects Med. 2005 Dec;26(6):459-516. doi: 10.1016/j.mam.2005.10.001. Epub 2005 Nov 23. PMID 16309738
- [Background] Ma L, Yan SF, Huang YM, Lu XR, Qian F, Pang HL, Xu XR, Zou ZY, Dong PC, Xiao X, Wang X, Sun TT, Dou HL, Lin XM. Effect of lutein and zeaxanthin on macular pigment and visual function in patients with early age-related macular degeneration. Ophthalmology. 2012 Nov;119(11):2290-7. doi: 10.1016/j.ophtha.2012.06.014. Epub 2012 Aug 1. PMID 22858124
- [Background] Piermarocchi S, Saviano S, Parisi V, Tedeschi M, Panozzo G, Scarpa G, Boschi G, Lo Giudice G; Carmis Study Group. Carotenoids in Age-related Maculopathy Italian Study (CARMIS): two-year results of a randomized study. Eur J Ophthalmol. 2012 Mar-Apr;22(2):216-25. doi: 10.5301/ejo.5000069. PMID 22009916
- [Background] Age-Related Eye Disease Study 2 Research Group. Lutein + zeaxanthin and omega-3 fatty acids for age-related macular degeneration: the Age-Related Eye Disease Study 2 (AREDS2) randomized clinical trial. JAMA. 2013 May 15;309(19):2005-15. doi: 10.1001/jama.2013.4997. PMID 23644932
- [Background] Trieschmann M, van Kuijk FJ, Alexander R, Hermans P, Luthert P, Bird AC, Pauleikhoff D. Macular pigment in the human retina: histological evaluation of localization and distribution. Eye (Lond). 2008 Jan;22(1):132-7. doi: 10.1038/sj.eye.6702780. Epub 2007 Mar 30. PMID 17401321
- [Background] Powner MB, Gillies MC, Tretiach M, Scott A, Guymer RH, Hageman GS, Fruttiger M. Perifoveal muller cell depletion in a case of macular telangiectasia type 2. Ophthalmology. 2010 Dec;117(12):2407-16. doi: 10.1016/j.ophtha.2010.04.001. Epub 2010 Aug 3. PMID 20678804
- [Background] Bone RA, Landrum JT, Fernandez L, Tarsis SL. Analysis of the macular pigment by HPLC: retinal distribution and age study. Invest Ophthalmol Vis Sci. 1988 Jun;29(6):843-9. PMID 3372161
- [Background] Morgan CL, Currie CJ, Stott NC, Smithers M, Butler CC, Peters JR. The prevalence of multiple diabetes-related complications. Diabet Med. 2000 Feb;17(2):146-51. doi: 10.1046/j.1464-5491.2000.00222.x. PMID 10746486
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Early photocoagulation for diabetic retinopathy. ETDRS report number 9. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):766-85. PMID 2062512
- [Background] Preliminary report on effects of photocoagulation therapy. The Diabetic Retinopathy Study Research Group. Am J Ophthalmol. 1976 Apr;81(4):383-96. doi: 10.1016/0002-9394(76)90292-0. PMID 944535
- [Background] Stefansson E. Ocular oxygenation and the treatment of diabetic retinopathy. Surv Ophthalmol. 2006 Jul-Aug;51(4):364-80. doi: 10.1016/j.survophthal.2006.04.005. PMID 16818083
- [Background] Mainster MA, Reichel E. Transpupillary thermotherapy for age-related macular degeneration: principles and techniques. Semin Ophthalmol. 2001 Jun;16(2):55-9. doi: 10.1076/soph.16.2.55.4213. PMID 15491004